CLINICAL TRIAL: NCT00236834
Title: A Multicenter, Randomized, Open Label Study to Compare the Safety and Efficacy of Levofloxacin With That of Imipenem/Cilastatin in the Treatment of Nosocomial Pneumonia
Brief Title: A Study of the Safety and Effectiveness of Levofloxacin Compared With Imipenem/Cilastatin in Patients With Pneumonia Acquired During Hospitalization
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Collaborators: PriCara, Unit of Ortho-McNeil, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR005557
Record Dates: First submitted 2005-10-07; First posted 2005-10-12 (Estimated); Last update posted 2011-06-10 (Estimated); Status verified 2010-04

CONDITIONS: Nosocomial Pneumonia
Keywords: respiratory tract diseases; levofloxacin; pneumonia; quinolones, hospital-acquired pneumonia; lung diseases
MeSH Terms: conditions — Healthcare-Associated Pneumonia; Respiratory Tract Diseases; Pneumonia; Lung Diseases | interventions — Levofloxacin; Imipenem

INTERVENTIONS:
Drug: levofloxacin; imipenem/cilastitin

SUMMARY:
The purpose of this study is to compare the safety and effectiveness of levofloxacin with imipenem/cilastatin in the treatment of hospital-acquired pneumonia

DETAILED DESCRIPTION:
Despite advances in prevention and treatment, hospital-acquired pneumonia remains a significant problem as the second most common infection acquired in the hospital and the most deadly (20%-50% of patients who acquire pneumonia while in the hospital die from complications of pneumonia). Levofloxacin has been shown in clinical trials to be effective against a number of different bacteria, including those found to be common and uncommon causes of pneumonia. This multicenter, open-label study evaluates the safety and effectiveness of levofloxacin as compared with imipenem/cilastatin, another type of antibiotic treatment, in patients with pneumonia acquired in the hospital. Patients receive treatment for a total of 7-15 days, initially with levofloxacin or imipenem/cilastatin, administered slowly through a vein. If patients respond positively to either drug, treatment may be changed to levofloxacin or ciprofloxacin (if initially treated with imipenem/cilastatin), to be taken by mouth. Certain additional drugs may be added if needed to treat pneumonia caused by certain bacteria. Patients showing signs of improvement continue in the study, with assessments 5-7 days (posttherapy visit) and 28-32 days after completion of the study drug (poststudy visit). Effectiveness is assessed by measuring the ability of the study drug to eliminate bacteria causing pneumonia and to reduce the signs and symptoms of pneumonia. Chest x-rays and laboratory tests for bacteria are performed throughout the study and patients' severity of disease is rated according to the Acute Physiology And Chronic Health Evaluation (APACHE) scale. Safety evaluations (incidence of adverse events, physical examinations, laboratory tests) are performed throughout the study. Blood samples are drawn from patients receiving levofloxacin to determine the concentration of levofloxacin in the blood. The study hypothesis is that levofloxacin is at least as effective as imipenem/cilastatin in treating hospital-acquired pneumonia and is generally well-tolerated.

Levofloxacin 750 mg administered through a vein once daily or imipenem/cilastatin 500mg-1 gram every 6-8 hours. Upon improvement, patients may transition to levofloxacin 750mg by mouth once daily or ciprofloxacin 750mg by mouth twice daily for 7-15 days.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of hospital-acquired pneumonia as follows: hospitalization >= 48 but <= 72 hours, identification of a bacteria commonly found in hospital-acquired infections, absence of pneumonia on initial chest x-ray, normal white blood cell count, and diagnosis other than infection upon admission to hospital OR hospitalized >= 72 hours OR discharged from a hospital <= 48 hours after a hospitalization of >= 72 hours AND chest x-ray findings consistent with infection AND abnormal temperature (high or low) or abnormal white blood cell count
* Specimen from respiratory tract is available for laboratory analysis
* APACHE score <= 35
* Have received at least 72 hours of treatment with antibiotics administered intravenously (through a vein) and have failed that treatment providing the previous drugs were not levofloxacin or imipenem/cilastatin and there is evidence of failure (specimen from respiratory tract documenting original bacteria causing pneumonia is still present or presence of a new bacteria causing pneumonia acquired in the hospital, continued abnormal temperature or worsening of x-ray findings and at least 1 of the following: increased white blood cell count or decrease in breathing ability/increase in oxygen requirements)
* Have received treatment with antibiotics administered intravenously (through a vein) for < 24 hours within 72 hours prior to study entry
* Hospitalized for >= 72 hours and develop acute signs and symptoms of pneumonia while on antibiotic(s) for another reason, providing that the previous antibiotic(s) were not levofloxacin or imipenem/cilastatin, no antibiotics have been given for the pneumonia and the previous antibiotic(s) can be discontinued

Exclusion Criteria:

* Infection due to a bacteria that is know to be resistant to levofloxacin or imipenem or certain other drugs that may be used during the study
* Have received treatment with antibiotics administered intravenously for > 24 hours within 72 hours prior to study entry
* Previous allergic or serious adverse reaction to any of the drugs used in this study or to a drug similar to those used in this study
* Cystic fibrosis or other lung disorder or an infection not treatable with antibiotics
* Significantly decreased kidney function
* Pre-infection terminal illness (such as cancer)
* Decreased white blood cell count

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 438 (Actual)
Dates: Start 1997-12; Study Completion 2001-06 (Actual)

PRIMARY OUTCOMES:
Microbiological response at posttherapy will be based on eradication or persistence of the pathogen(s) isolated at admission

SECONDARY OUTCOMES:
Clinical response at posttherapy will be based on the comparison of posttherapy signs/symptoms and radiological findings reported at posttherapy compared to those reported at admission. Clinical and microbiologic response at poststudy.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research and Development, L.L.C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- [Result] West M, Boulanger BR, Fogarty C, Tennenberg A, Wiesinger B, Oross M, Wu SC, Fowler C, Morgan N, Kahn JB. Levofloxacin compared with imipenem/cilastatin followed by ciprofloxacin in adult patients with nosocomial pneumonia: a multicenter, prospective, randomized, open-label study. Clin Ther. 2003 Feb;25(2):485-506. doi: 10.1016/s0149-2918(03)80091-7. PMID 12749509
- See also: A study of the safety and effectiveness of levofloxacin compared with imipenem/cilastatin in patients with pneumonia acquired during hospitalization — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=664&filename=CR005557_CSR.pdf